CLINICAL TRIAL: NCT06412679
Title: Rebuilding Emotional Stability and Strength Through Therapeutic and Life-Skills Education for Internally Displaced Persons in Nigeria (RESETTLE-IDPs): a Hybrid Type II Effectiveness-implementation Study
Brief Title: RESETTLE-IDPs: Life-Skills Education and Psychosocial Resilience Building for Displaced Nigerians
Acronym: RESETTLE-IDPs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: University of Maiduguri Teaching Hospital (Unknown); Brooks Insights Limited (Unknown)
Responsible Party: Principal Investigator, Ejemai Eboreime, Assistant Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-7085; PAA - 192178 (Other Grant/Funding Number: CIHR); R-HGC-POC-2408-67370 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Mental Health; Psychosocial Functioning; Implementation Science; Global Health; Conflict
Keywords: Conflict; Forced Displacement; Internally displaced persons; Mental health; Psychosocial support; Life skills education; Mobile health; Digital health; Humanitarian emergencies; Global mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Type II Hybrid Effectiveness-Implementation Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-Person Life Skills Education (LSE) Peer Support Groups (Active Comparator): Participants will receive a culturally-adapted LSE intervention delivered through weekly in-person peer support group sessions for 12 weeks. The LSE curriculum covers topics such as stress management, communication skills, problem-solving, emotion regulation, health and hygiene, social skills, gender norms and safety, education and livelihoods, and community mobilization. Each peer support group will consist of 10-12 participants, separated by gender and age bands (12-17 and 18-24 for youth, 18+ for women), and will meet weekly for approximately 2 hours in a private, safe space within the IDP camp. Sessions will be co-facilitated by a trained IDP peer leader and a local mental health provider, following a structured format with interactive activities, discussions, and skill practice.
  Interventions: Behavioral: Life Skills Education
- WhatsApp-Enabled LSE Virtual Peer Support Groups (Active Comparator): Participants will receive the same culturally-adapted LSE curriculum as those in the In-person arm, but delivered through WhatsApp for 12 weeks. Participants will be added to a moderated WhatsApp group chat with other IDP youth or women in their camp, where they will receive three LSE-related messages per week. These messages will include brief psychoeducational content, practice exercises, reflection prompts, and reminders to engage with the virtual support group. The WhatsApp group will provide a platform for participants to discuss the LSE topics, share experiences and coping strategies, and provide emotional support to one another, with trained IDP peer facilitators moderating the chats to ensure a safe and supportive environment. Participants will also receive regular push notifications with motivational messages, links to further resources, and reminders to practice the LSE skills.
  Interventions: Behavioral: Life Skills Education

INTERVENTIONS:
Behavioral: Life Skills Education — The RESETTLE-IDPs study compares two innovative delivery approaches for a culturally-adapted life skills education (LSE) intervention aimed at improving the mental health and well-being of internally displaced persons in Nigeria. The interventions are distinguished by their mode of delivery (in-person vs. WhatsApp-based), their focus on peer support and skill-building, and their tailoring to the specific needs and challenges of IDP populations.

SUMMARY:
The RESETTLE-IDPs study aims to address the urgent mental health needs of internally displaced youth and women in Nigeria, who face high rates of depression, anxiety, and post-traumatic stress due to exposure to conflict, violence, and loss. Despite the immense needs, there is a severe lack of culturally appropriate, evidence-based interventions to support the resilience and well-being of these vulnerable populations.

To fill this gap, the study will evaluate the effectiveness and implementation of a novel life skills education (LSE) program delivered through two innovative approaches: in-person peer support groups and WhatsApp-based virtual support groups. The LSE curriculum, developed through extensive community engagement, covers topics such as stress management, communication, problem-solving, health, safety, and advocacy, all tailored to the unique challenges of displacement.

In the in-person arm, trained IDP peers and local providers will facilitate weekly group sessions over 12 weeks, providing a safe space for participants to learn, practice, and apply new skills while building social connections and support networks. In the WhatsApp arm, participants will receive weekly messages with educational content, reflection prompts, and exercises, moderated by trained facilitators to foster dialogue and peer support.

By comparing these two delivery methods, the study aims to identify the most feasible, acceptable, and effective strategies for rolling out psychosocial support interventions in humanitarian settings, particularly those with limited resources and access. The study will also assess the interventions' impact on key mental health outcomes, including depression, anxiety, PTSD, and well-being, as well as life skills, functioning, and implementation metrics such as reach, adoption, and sustainability.

Ultimately, the RESETTLE-IDPs study seeks to generate actionable evidence to inform the development and scale-up of culturally responsive, community-driven interventions that can promote the mental health and resilience of conflict-affected populations in Nigeria and beyond. By empowering IDP youth and women with the knowledge, skills, and support to navigate the challenges of displacement, the study aims to contribute to a brighter, more hopeful future for these resilient communities

DETAILED DESCRIPTION:
The RESETTLE-IDPs study is a cluster-randomized type II effectiveness-implementation hybrid trial that aims to evaluate the effectiveness and implementation of a life skills education (LSE) intervention delivered through two innovative approaches - in-person peer support groups and WhatsApp-based virtual support groups - to improve the mental health and well-being of internally displaced persons in Nigeria.

Background and Rationale:

Nigeria is facing a severe humanitarian crisis, with over 2.7 million people internally displaced due to armed conflict, communal violence, and natural disasters. Internally displaced persons (IDPs) in Nigeria, particularly youth and women, are at high risk of mental health problems such as depression, anxiety, and post-traumatic stress disorder (PTSD) due to exposure to trauma, loss, and ongoing stressors. Despite the immense needs, there is a severe lack of culturally appropriate, evidence-based interventions to support the mental health and resilience of IDP populations in Nigeria and other low-resource humanitarian settings.

Life skills education (LSE) is a promising approach to promoting mental health and well-being among conflict-affected populations. LSE programs aim to equip individuals with the knowledge, attitudes, and skills needed to navigate challenges, cope with stress, and make healthy decisions. Previous studies have shown that LSE interventions can improve mental health outcomes, social-emotional learning, and positive youth development in various contexts. However, there is limited evidence on the effectiveness and implementation of LSE programs specifically tailored for IDP youth and women in Nigeria, and how different delivery methods (e.g., in-person vs. mobile-based) may impact their reach, acceptability, and sustainability.

Study Objectives:

The primary objective of the RESETTLE-IDPs study is to evaluate the effectiveness of a 12-week LSE intervention, delivered through either in-person peer support groups or WhatsApp-based virtual support groups, on mental health outcomes (depression, anxiety, PTSD, and well-being) among IDP youth and women in Nigeria, compared to a wait-list control group.

Secondary objectives include:

1. To assess the impact of the LSE intervention on life skills acquisition, daily functioning, and social support among IDP youth and women.
2. To compare the feasibility, acceptability, fidelity, and cost-effectiveness of in-person vs. WhatsApp-based delivery methods for the LSE intervention.
3. To explore the contextual factors, implementation processes, and mechanisms of change that influence the effectiveness and sustainability of the LSE intervention in IDP settings.
4. To engage stakeholders (IDP communities, health workers, humanitarian organizations, policymakers) in the design, implementation, and evaluation of the LSE intervention to promote its cultural relevance, ownership, and scalability.

Methods: The study will use a three-arm cluster-randomized controlled trial design, with IDP camps in Nigeria randomly allocated to one of two groups: (1) in-person LSE peer support groups, (2) WhatsApp-based LSE virtual support groups. The target population includes IDPs youth aged 13 years and above residing in selected camps in Borno State, the epicenter of the Boko Haram insurgency and displacement crisis in Nigeria.

The intervention will consist of a culturally adapted LSE curriculum covering topics such as stress management, communication skills, problem-solving, health and hygiene, safety and protection, gender norms, and community mobilization. The curriculum will be developed through a participatory process involving IDP youth and women, community leaders, health workers, and education specialists, drawing on existing evidence-based resources and guidelines (e.g. UNICEF LSE Toolkit).

In the in-person arm, trained IDP peers and local providers will facilitate weekly gender- and age-segregated support groups of 10-12 participants over a 12-week period. The groups will provide a safe space for participants to learn and practice life skills, share experiences, and provide mutual support. Sessions will use interactive, experiential learning methods such as role-plays, discussions, and group projects.

In the WhatsApp arm, participants will be enrolled in moderated virtual support groups that deliver the LSE curriculum through weekly conversations, including psychoeducational content, reflection prompts, skill-building exercises, and peer discussion topics. Trained IDP facilitators will moderate the groups to ensure safe and supportive interactions, provide feedback, and encourage skill application.

The study will enroll a total of 500 participants (250 per arm) across 20 IDP camps, with an estimated 25 participants per camp. Participants will be recruited through community-based mobilization strategies, with support from camp leaders, health workers, and NGO partners.

Data will be collected at baseline, 3 months, 6 months, and 12 months using a combination of quantitative and qualitative methods. Quantitative data will include validated mental health scales, as well as locally adapted measures of life skills, functioning, and social support. Qualitative data will include in-depth interviews and focus group discussions with participants, facilitators, and stakeholders to explore experiences, perceptions, and contextual factors influencing the intervention.

Data analysis will use an intent-to-treat approach, with mixed-effects regression models to assess intervention effects on primary and secondary outcomes, accounting for clustering at the camp level. Qualitative data will be analyzed thematically to identify barriers, facilitators, and mechanisms of change. Implementation outcomes (e.g., reach, fidelity, acceptability) will be assessed using process evaluation frameworks (e.g., RE-AIM).

Expected Results and Impact:

The RESETTLE-IDPs study aims to generate rigorous evidence on the effectiveness and implementation of a culturally adapted LSE intervention for improving the mental health and well-being of IDP youth and women in Nigeria. The study findings will have important implications for the design, delivery, and scale-up of psychosocial support interventions in humanitarian settings, particularly those affected by conflict and displacement.

By comparing in-person and WhatsApp-based delivery methods, the study will provide valuable insights into the relative advantages, challenges, and effectiveness of different approaches to reaching and engaging IDP populations. The use of implementation science frameworks and participatory research methods will ensure that the intervention is not only effective but also feasible, acceptable, and sustainable in real-world contexts.

The study will also contribute to capacity-building and empowerment of IDP communities by training and engaging youth and women as peer facilitators, researchers, and advocates. The participatory approach aims to foster local ownership, leadership, and sustainability of the intervention beyond the research period.

Ultimately, the RESETTLE-IDPs study has the potential to inform policy, practice, and funding priorities for mental health and psychosocial support in humanitarian settings, both in Nigeria and globally. By advancing the evidence base on culturally relevant, community-based interventions, the study can contribute to reducing the global burden of mental health disorders and promoting the resilience and well-being of conflict-affected populations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 years and above
* Ownership of smartphone
* Internally displaced for at least 6 months.
* Residing in select IDP camps in Abuja and Borno State, Nigeria
* Fluency in English and/or Hausa languages
* Willing and able to provide informed consent.

Exclusion Criteria:

* Active suicidal ideation or attempts (i.e having thoughts, plans, or intent to end one's life within the past month)
* Active psychosis
* Cognitive impairment precluding informed consent or survey completion.
* Not owning as smartphone

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Post-Traumatic Stress Disorder (PTSD) symptoms | Baseline, 3 months, 6 months, and 12 months
  Metric/Method of Measurement: PTSD Checklist for DSM-5 (PCL-5) The PCL-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms based on the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria. Participants rate how much they have been bothered by each symptom in the past month on a 5-point scale ranging from 0 (not at all) to 4 (extremely). The total score ranges from 0 to 80, with higher scores indicating greater severity of PTSD symptoms. A score of 31-33 or higher suggests probable PTSD diagnosis.

SECONDARY OUTCOMES:
Change in depressive symptoms | Baseline, 3 months, 6 months, and 12 months
  Metric/Method of Measurement: Patient Health Questionnaire-9 (PHQ-9) The PHQ-9 is a 9-item self-report measure that assesses the presence and severity of depressive symptoms based on the DSM-5 criteria. Participants rate how often they have been bothered by each symptom over the past 2 weeks on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms. Cut-off scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively.
Change in anxiety symptoms | Baseline, 3 months, 6 months, and 12 months
  Metric/Method of Measurement: Generalized Anxiety Disorder-7 (GAD-7) The GAD-7 is a 7-item self-report measure that assesses the presence and severity of anxiety symptoms. Participants rate how often they have been bothered by each symptom over the past 2 weeks on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21, with higher scores indicating greater severity of anxiety symptoms. Cut-off scores of 5, 10, and 15 represent mild, moderate, and severe anxiety, respectively.
Change in life skills | Baseline, 3 months, 6 months, and 12 months
  Metric/Method of Measurement: A Life Skills Assessment Tool (LSAT) The LSAT is a locally developed measure that assesses participants' knowledge, attitudes, and behaviors related to the key life skills covered in the LSE curriculum (e.g., stress management, communication, problem-solving, health and hygiene). The scale includes a mix of multiple-choice and Likert-type items, with higher scores indicating greater life skills competency. The exact number of items and scoring system will be determined through formative research and pilot testing with the target population.
Change in well-being | Baseline, 3 months, 6 months, and 12 months
  Metric/Method of Measurement: World Health Organization-Five Well-Being Index (WHO-5) The WHO-5 is a 5-item self-report measure that assesses subjective psychological well-being over the past 2 weeks. Participants rate each item on a 6-point scale ranging from 0 (at no time) to 5 (all of the time). The total score ranges from 0 to 25, which is then multiplied by 4 to yield a percentage score ranging from 0 to 100. A score below 50 suggests poor well-being and a score below 28 indicates likely depression.
Change in perceived appropriateness of the intervention | Baseline, 3 months
  Metric/Method of Measurement: Intervention Appropriateness Measure (IAM) The IAM is a 4-item self-report measure that assesses the perceived appropriateness of an intervention. Participants rate each item on a 5-point scale ranging from 1 (completely disagree) to 5 (completely agree). The total score ranges from 4 to 20, with higher scores indicating greater appropriateness.
Change in acceptability of the intervention | Baseline, 3 months
  Metric/Method of Measurement: Acceptability of Intervention Measure (AIM) The AIM is a 4-item self-report measure that assesses the perceived acceptability of an intervention. Participants rate each item on a 5-point scale ranging from 1 (completely disagree) to 5 (completely agree). The total score ranges from 4 to 20, with higher scores indicating greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Ejemai A Eboreime, MBBS, PhD, Principal Investigator — Dalhousie University; Vincent Agyapong, MD, PhD, Principal Investigator — Dalhousie University; Rita Orji, PhD, Principal Investigator — Dalhousie University; Sanni Yaya, PhD, Principal Investigator — University of Ottawa
Locations (1):
- Wassa and Durumi IDP camps, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified IPD underlying the published results of the RESETTLE-IDPs study, including the study protocol, statistical analysis plan, and analytic code.
  IPD will be made available upon reasonable request and after approval by the study's steering committee, subject to a data sharing agreement
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Data Sharing Statement We will share de-identified IPD underlying the published results of the RESETTLE-IDPs study, including the study protocol, statistical analysis plan, and analytic code.
  IPD will be made available upon reasonable request and after approval by the study's steering committee, subject to a data sharing agreement.
  Access Criteria and Procedure Researchers interested in accessing the IPD should submit a formal request to the study's principal investigator, specifying the purpose, scope, and timeline of the proposed analyses.
  Requests will be reviewed by the steering committee based on the scientific merit, feasibility, and alignment with the study's objectives and participants' informed consent.
URL: ftp://NA

REFERENCES:
- [Background] Kaiser BN, Ticao C, Boglosa J, Minto J, Chikwiramadara C, Tucker M, Kohrt BA. Mental health and psychosocial support needs among people displaced by Boko Haram in Nigeria. Glob Public Health. 2020 Mar;15(3):358-371. doi: 10.1080/17441692.2019.1665082. Epub 2019 Sep 19. PMID 31535595
- [Background] Ugbe UM, Esu EB, Efut JA, Bisongedam MM, Awa TM, Ekpo OI. Sociodemographic correlates and associated factors of depression and anxiety among internally displaced adults in Ogoja, Nigeria. Gen Psychiatr. 2022 Apr 28;35(2):e100749. doi: 10.1136/gpsych-2022-100749. eCollection 2022. PMID 35572773
- [Background] Wei Y, Hayden JA, Kutcher S, Zygmunt A, McGrath P. The effectiveness of school mental health literacy programs to address knowledge, attitudes and help seeking among youth. Early Interv Psychiatry. 2013 May;7(2):109-21. doi: 10.1111/eip.12010. Epub 2013 Jan 24. PMID 23343220
- [Background] Taubner S, Ioannou Y, Saliba A, Sales CMD, Volkert J, Protic S, Adler A, Barkauskiene R, Conejo-Ceron S, Di Giacomo D, Mestre JM, Moreno-Peral P, Vieira FM, Mota CP, Henriques MIRS, Rossberg JI, Perdih TS, Schmidt SJ, Zettl M, Ulberg R, Heinonen E. Mediators of outcome in adolescent psychotherapy and their implications for theories and mechanisms of change: a systematic review. Eur Child Adolesc Psychiatry. 2024 Oct;33(10):3321-3358. doi: 10.1007/s00787-023-02186-9. Epub 2023 Mar 15. PMID 36918434
- [Background] Sahebalzamani M, Farahani H, Feizi F. Efficacy of life skills training on general health in students. Iran J Nurs Midwifery Res. 2012 Nov;17(7):553-5. PMID 23922605
- [Background] Singla DR, Waqas A, Hamdani SU, Suleman N, Zafar SW, Zill-E-Huma, Saeed K, Servili C, Rahman A. Implementation and effectiveness of adolescent life skills programs in low- and middle-income countries: A critical review and meta-analysis. Behav Res Ther. 2020 Jul;130:103402. doi: 10.1016/j.brat.2019.04.010. Epub 2019 Apr 26. PMID 31146889
- [Background] Maghsoudi J, Sabour NH, Yazdani M, Mehrabi T. The effect of acquiring life skills through humor on social adjustment rate of the female students. Iran J Nurs Midwifery Res. 2010 Fall;15(4):195-201. PMID 22049280
- [Background] Magnani R, Macintyre K, Karim AM, Brown L, Hutchinson P, Kaufman C, Rutenburg N, Hallman K, May J, Dallimore A; Transitions Study Team. The impact of life skills education on adolescent sexual risk behaviors in KwaZulu-Natal, South Africa. J Adolesc Health. 2005 Apr;36(4):289-304. doi: 10.1016/j.jadohealth.2004.02.025. PMID 15780784
- [Background] undefined
- [Derived] Eboreime E, Obi-Jeff C, Orji R, Ojo TM, Iyamu I, Harri BI, Said JM, Oguntimehin F, Ibrahim A, Anjorin O, Duke AEE, Musami UB, Liebenberg L, Crider R, Wagami L, Dahiru AM, Uneke JC, Yaya S, Agyapong VI. In-person vs mobile app facilitated life skills education to improve the mental health of internally displaced persons in Nigeria: protocol for the RESETTLE-IDPs cluster randomized hybrid type 2 effectiveness-implementation trial. BMC Health Serv Res. 2024 Oct 22;24(1):1269. doi: 10.1186/s12913-024-11762-x. PMID 39438885